CLINICAL TRIAL: NCT02461901
Title: Does Using Fidaxomicin to Treat Clostridium Difficile Infection (CDI) Reduce the Recovery of C. Difficile From Patients' Faeces, Skin and Their Immediate Environment, Compared to Treatment With Vancomycin or Metronidazole?
Brief Title: Does Fidaxomicin Therapy Reduce Spread of Clostridium Difficile?
Status: Completed | Type: Observational
Sponsor: Professor Mark Wilcox (Other)
Collaborators: Astellas Pharma Europe Ltd. (Industry); The Leeds Teaching Hospitals NHS Trust (Other); St George's Healthcare NHS Trust (Other)
Responsible Party: Sponsor-Investigator, Professor Mark Wilcox, Professor of Medical Microbiology, University of Leeds
Organization: University of Leeds (Other)
Other Study IDs: 14/NW/1398
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Clostridium Difficile Infection
Keywords: clostridium difficile; environment; contamination; fidaxomicin
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Isolates of Clostridium difficile
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fidaxomicin treatment: Patients being treat with fidaxomicin (on the decision of their treating physician)
  Interventions: Other: Environmental sampling; Other: Skin swab sampling; Other: Fecal sampling
- Metronidazole or vancomycin treatment: Patients being treated with metronidazole or vancomycin (on the decision of their treating physician)
  Interventions: Other: Environmental sampling; Other: Skin swab sampling; Other: Fecal sampling

INTERVENTIONS:
Other: Environmental sampling — Sampling of five sites in the patient's immediate environment for C. difficile spores
Other: Skin swab sampling — Collection of swabs from three sites on the skin for C. difficile spores
Other: Fecal sampling — Collection of fecal samples for C. difficile spores

SUMMARY:
This study evaluates whether patients with Clostridium difficile infection (CDI) who are treated with fidaxomicin have less contamination of their skin and surrounding environment with spores of C. difficile than patients treated with other drugs (metronidazole or vancomycin)

DETAILED DESCRIPTION:
Fidaxomicin is a newly licensed drug for the treatment of CDI. Patients treated with fidaxomicin have a significantly lower C. difficile spore count in their faeces than patients who receive alternative drugs (metronidazole or vancomycin). In vitro evidence has shown that the drug persists in the gut for several weeks after treatment has finished and also prevents the outgrowth of spores. These findings suggest that fidaxomicin therapy could be associated with less contamination of CDI patient's skin and their surrounding environment than metronidazole or vancomycin therapy.

This prospective, case control study aims to investigate this hypothesis by measuring C. difficile spore counts in patient's stool samples, on their skin and in the surrounding environment. Results for patients receiving fidaxomicin will be compared with those on either metronidazole or vancomycin.

If fidaxomicin therapy does reduce contamination levels, it might be a useful adjunct to existing measures used to control CDI in healthcare settings, particularly in outbreak situations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CDI (see above)
* Prescribed fidaxomicin, vancomycin or metronidazole by attending physician

Exclusion Criteria:

* Patients whose clinical care team indicates it would be inappropriate to include him/her in the study (e.g. due to terminal illness)
* In a patient receiving metronidazole or vancomycin, receipt of fidaxomicin within the previous 3 months
* patients unable to give informed consent for whom no consultee is available to give approval
* non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Clostridium difficile infection.
  CDI is defined as the presence of both:
  * a positive C. difficile toxin assay result on a fecal sample, and
  * diarrhea (Bristol stool type 5-7) >/= 3 times in any 24 hour period in the last 7 days
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12-31 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The presence of environmental contamination with C. difficile spores during and following treatment with fidaxomicin, vancomycin or metronidazole. | Up to 28 days after treatment
The presence of skin contamination with C. difficile spores during and following treatment with fidaxomicin, vancomycin or metronidazole. | Up to 28 days after treatment

SECONDARY OUTCOMES:
C.difficile spore counts in the faeces of CDI patients before, during and after treatment with fidaxomicin, vancomycin or metronidazole. | Up to 28 days after treatment
Total C. difficile spore counts from skin swab samples during and following treatment with fidaxomicin, vancomycin or metronidazole. | Up to 28 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Wilcox, Study Chair — Leeds Teaching Hospitals NHS Trust; Tim Planche, Principal Investigator — St George's Healthcare NHS Trust; Philip Stanley, Principal Investigator — Bradford Teaching Hospitals NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - St George's University Hospitals NHS Foundation Trust, Tooting, London
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Undecided